CLINICAL TRIAL: NCT04702646
Title: Agreement Between Cleansing Quality Assessment During Colonoscopy and Patient Reported Cleansing Quality
Brief Title: Patient and Colonoscopy Cleansing Quality Agreement
Acronym: CALPER
Status: Completed | Type: Observational
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Other Study IDs: Colon cleansing agreement
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cleansing Quality of the Colon
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive patients for outpatient colonoscopy: The researchers will offer to participate in the study to patients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria
  Interventions: Drug: Bowel preparation before colonoscopy; Procedure: Colonoscopy

INTERVENTIONS:
Drug: Bowel preparation before colonoscopy — one day liquid diet will be administered to every patient included in the study and: split-dose bowel preparation with 4 Liters of Polyethylene glycol solution, 2 Liters of PEG-Ascorbic acid or 2 Liters Picosulfate.
Procedure: Colonoscopy — colonoscopy will be performed to every patient included in the study

SUMMARY:
The main purpose of the study is to determine the agreement between colon cleansing quality assessed by a validated scale (Boston Bowel Preparation Scale, BBPS) and the perception of the patient. Patients will be prepared with polyethylene glycol (PEG), PEG plus ascorbic acid (PEG-Asc) or sodium picosulfate-oxide magnesium solution (PS).

The secondary aim is to assess predictors of poor bowel cleansing.

DETAILED DESCRIPTION:
Although, current guidelines recommend a rate of inadequate bowel cleansing for colonoscopy not higher than 10-15%, in clinical practice poor bowel cleansing in endoscopy units ranged between 6.8% and 33 The patient's perception of their colon cleansing before colonoscopy has been stated as a predictor of cleansing quality in a limited number of studies. In such a way, if the agreement between the patient's reported colon cleansing and the quality during colonoscopy is optimal, rescue cleansing strategies such as the administration of additional bowel solution might be indicated. In the studies that assessed the relationship between patient and colonoscopy assessment of colon cleansing quality the agreement was fair. The main drawback of these studies is that they do not used a validated colonoscopy cleansing scale.

Therefore, ideally, patient-referred information regarding the quality of colon cleaning could be a factor of great value in guiding rescue strategies. However, the available evidence of the correlation between the patient's perception of the quality of colon cleansing at the time of colonoscopy is scarce and has also not been adequately studied. Evaluating this correlation in a cohort of unselected patients referred for outpatient colonoscopy and using a universally accepted validated colon cleansing quality scale could help to determine whether this system is a good predictor of inadequate colon cleansing and can guide the implementation of rescue strategies.

The researchers will offer to participate in the study to patients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information. Patients will fill out a questionnaire on the day of colonoscopy on the perception of cleanliness based on the last stool. To do this, a set with 4 figures (light liquid, light liquid with lumps, dark liquid or solid particles) used in a previous study will be shown to the patient and the patient should indicate which figure is more similar to the last bowel movement. Optionally, the patient will be able to provide the investigating staff with a photo of their last deposition. Patients should also note the hour of the last stool. Four researchers will chose the set considered more appropriate for the study.

In addition, three sets compound of 4 pictures of different cleansing qualities will be presented to a subgroup of patients to test which one is more similar to the last stool.

Subsequently, the colonoscopy will be performed and the cleaning quality will be scored according to the BBPS considering suboptimal a cleaning quality of less than 2 points in a segment of the colon. Patients will receive any of the routinely used colonic preparations in the hospital, i.e. Casenglycol® (polyethylene glycol), Moviprep® (polyethylene glycol and ascorbic acid) and Citrafleet® (picosulfate sodium, light magnesium oxide, citric acid).The bowel cleansing quality following BBPS will be assessed by the endoscopist.

The aim of this study is to test the agreement between the colon cleansing quality assessed by the BBPS and the patient reported colon quality.

In our unit the percentage of colonoscopies with poor preparation in unselected population is about 15-20% of patients undergoing colonoscopy. For the logistic regression model it is necessary to include 10 patients with poor preparation for each variable. Initially hypothesizing that we will include 9 variables, a total of 600 patients will be required.

The t Student test will be used to compare groups in continuous variables. All values of p <0.05 shall be considered significant.

A univariate analysis will be performed comparing each of the possible predictor variables with the dependent variable with the cleaning quality during colonoscopy (BBPS ≥ 2 in each segment). Subsequently, a logistic regression analysis will be carried out to evaluate the predictor factors of adequate quality evaluated by the BBPS including those with a significance of ≤ 0.15.

ELIGIBILITY:
Inclusion Criteria:

* Age >18,
* to sign the informed consent
* patients with indication of outpatient colonoscopy
* patient ingesting preparation

Exclusion Criteria:

* Last colonoscopy with poor bowel preparation.
* Ileus, intestinal obstruction, megacolon.
* Poorly controlled hypertension (systolic hypertension> 180mmHg, dyastolic hypertension> 100mmHg).
* Terminal renal failure (pre-dialysis or dialysis).
* Congestive heart failure (NYHA III-IV).
* Acute liver failure.
* Severe psychiatric illness.
* Dementia with difficulty in the intake of the preparation.
* Pregnancy or breastfeeding.
* Refusal to participate in the study.
* Allergies.
* Not looking at the characteristics of the last stool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researchers will offer to participate in the study to patients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information.
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of bowel cleansing | [Time frame: 1 years][Designated as safety issue: No]
  Quality of bowel cleansing assessed by the Boston Bowel Preparation Scale. This scale goes from 0 (no preparation) to 3 points (excellent preparation) in the three segments of the colon (proximal, transverse and distal). The maximum score is 9 points

SECONDARY OUTCOMES:
Predictive factors associated to an adequate bowel cleansing | [Time Frame: 1 years][Designated as safety issue: No]
  Predictive factors of poor bowel preparation will be evaluated in a logistic regression analysis
Test the correlation between 3 sets of pictures and the cleansing quality following the Boston Bowel Preparation Scale | [Time Frame: 6 months][Designated as safety issue: No]
  Three sets of 4 different quality pictures will be presented to the patients. Patients should choose the picture more similar to the last stool of each set.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z Gimeno Garcia, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Department of Gastroenterology, San Cristóbal de La Laguna, S/C de Tenerife, Spain

REFERENCES:
- [Background] Fatima H, Johnson CS, Rex DK. Patients' description of rectal effluent and quality of bowel preparation at colonoscopy. Gastrointest Endosc. 2010 Jun;71(7):1244-1252.e2. doi: 10.1016/j.gie.2009.11.053. Epub 2010 Apr 1. PMID 20362286
- [Background] Harewood GC, Wright CA, Baron TH. Assessment of patients' perceptions of bowel preparation quality at colonoscopy. Am J Gastroenterol. 2004 May;99(5):839-43. doi: 10.1111/j.1572-0241.2004.04176.x. PMID 15128347
- [Background] ASGE Technology Committee; Mamula P, Adler DG, Conway JD, Diehl DL, Farraye FA, Kantsevoy SV, Kaul V, Kethu SR, Kwon RS, Rodriguez SA, Tierney WM. Colonoscopy preparation. Gastrointest Endosc. 2009 Jun;69(7):1201-9. doi: 10.1016/j.gie.2009.01.035. No abstract available. PMID 19481646
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Background] Hernandez G, Gimeno-Garcia AZ, Quintero E. Strategies to Improve Inadequate Bowel Preparation for Colonoscopy. Front Med (Lausanne). 2019 Nov 8;6:245. doi: 10.3389/fmed.2019.00245. eCollection 2019. PMID 31781565